CLINICAL TRIAL: NCT06409598
Title: Efficacy of NOn-immersive Virtual Reality Adapted Telerehabilitation Exercises for Upper Limb Function and Balance (NOVEL) Program in Stroke Patients: A Mixed Method Pilot Feasibility Study.
Brief Title: NOVEL Program for Stroke Telerehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Stroke Telerehabilitation
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Chronic Stroke
Keywords: virtual reality; Telerehabilitation; Qualitative; Feasibility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded from knowing if the participant assigned to the experimental or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-immersive virtual reality intervention (Experimental): The experimental group will receive the NOVEL (NOn-immersive Virtual reality Exercises for for upper Limb function and balance) program. This adapted program consists of 4 different non-immersive home-based virtual reality exercise games tailored for upper limb and static balance training combined with motivational strategies (performance feedback, automated progression, exercise gamification) and previously used with non-stroke populations. A videoconferencing or phone call session will be done with the main researcher once per week (Asynchronous with the sessions) to check for any technical difficulties, monitor the progression of the exercises and the progression of the difficulty levels).
  Dose of exercises: the participant will have to use the exercise platforms for a minimum of 1 hour per day for 5 days per week. The total period of the intervention will be 8 weeks.
  Interventions: Other: Non-immersive virtual reality home-based exercise.
- Usual care (No Intervention): Stroke survivors assigned to the control group will continue to receive their usual care in accordance with local policies and practices. Usually, there is no available formal rehabilitation protocol for stroke survivors in the chronic stage of their recovery , but they are considered for long-term management and secondary prevention. No attempt will be made to discourage the provision of additional care, to ensure that usual care is provided. As part of the usual care trial, patients' activity records will be monitored by the researcher, in order to record any stroke care that can be provided to the patients during the trial period.

INTERVENTIONS:
Other: Non-immersive virtual reality home-based exercise. — This intervention aims include some exercises in the form of games to facilitate and improve the upper limb functions and static balance from sitting and standing positions among chronic stroke survivors.
  Arms: Non-immersive virtual reality intervention

SUMMARY:
Strokes are estimated to be the third most common cause of death in the world and the second most common cause of disability. Recently, the incidence of stroke has increased due to population aging. It is common for stroke survivors to experience a functional decline in their capacity to carry out daily activities as a consequence of their increasing dependence, which ultimately affects motivation levels, self-efficacy, and quality of life. Following a stroke, people often experience problems with upper limb function. Over half of people with upper limb impairments who have suffered a stroke continue to experience problems months or years afterward.

A significant amount of rehabilitation is necessary to obtain meaningful recovery in the upper extremities and balance, but such interventions are difficult to access.

As a cutting-edge method of neurorehabilitation, extended reality technology like virtual reality provides a more intensive simulation of functional activities than traditional physical therapy methods (aerobic, resistance, flexibility exercises, balance and coordination training, and functional exercises. The non-immersive type of VR can provide the patient with a safe experience so they can practice their exercises using gamification features integrated into the VR system, while remaining aware of their surroundings.

According to the most recently published studies, there is promising evidence regarding the use of home-based exercises in stroke management especially after the Covid-19 pandemic. However, there is still a gap in identifying the evidence for using non-immersive home-based virtual reality exercises as telerehabilitation on the upper limb function and balance motor outcomes, adherence, and compliance with rehabilitation programs. In addition, no study have evaluated the validity and fidelity of the gamified features that can be added to the non-immersive VR exercises in terms of improving patient adherence and experience to their rehabilitation program. Moreover, the investigators still need rigorous qualitative studies to explore patient experiences after doing these exercises at home with remote monitoring from their rehabilitation team.

DETAILED DESCRIPTION:
Physical recovery from stroke requires very large numbers of high-quality repetitive, task-directed movements, conventionally delivered face-to-face by therapists and assistants. Stroke is the single largest cause of complex disability in the UK [NHS LTP]. Around 100,000 people have a stroke in the UK each year and there are currently about 1.2 million UK stroke survivors. The annual UK cost of formal social care for people with stroke in 2015 was estimated at £5.2 billion and is expected to more than triple by 2035. Strokes are estimated to be the third most common cause of death in the world and the second most common cause of disability. Recently, the incidence of stroke has increased due to population aging. It is common for stroke survivors to experience a functional decline in their capacity to carry out daily activities as a consequence of their increasing dependence, which ultimately affects motivation levels, self-efficacy, and quality of life.

Following a stroke, people often experience problems with upper limb function. Over half of people with upper limb impairments who have suffered a stroke continue to experience problems months or years afterward. A common symptom of these upper limb impairments is difficulty moving and coordinating the arms, hands, and fingers, which may make it challenging to carry out daily tasks such as eating, dressing, and cleaning. Enhancing arm function is, therefore, an essential component of rehabilitation. An array of possible interventions have been developed, including different exercises or training, specialist equipment or techniques (splints), or the use of a drug to facilitate arm movement (Botox injections).

In stroke patients, balance impairment is one of the biggest obstacles to independence. Balance could be classified into static balance and dynamic balance. Many peope with stroke experience reduced balance due to deficits in motor control. Maintaining an upright posture to maintain balance requires good motor control; poor postural control adversely affects balance. In stroke patients, decreased static and dynamic balance poses a significant risk for falls and limits their ability to perform daily tasks. Therefore, restoring functional balance is one of the main goals of stroke rehabilitation, and restoring proper postural control is essential in order to be able to carry out daily living activities independently.

A significant amount of rehabilitation is necessary to obtain meaningful recovery in the upper extremities and balance, but such interventions are difficult to access. Inpatient rehabilitation is generally only permitted for a short period of time, and outpatient rehabilitation is limited in duration. Accordingly, home-based rehabilitation plays a crucial role in the rehabilitation continuum, allowing continuous and sufficient rehabilitation over a prolonged period of time, thereby improving function. Home-based rehabilitation or self-training are also important considering patients' mobility issues, transportation problems, or caregiver issues when trying to access rehabilitation facilities.

Its virtual environment provides users with the opportunity to learn and practice their exercise in a highly motivating and adherence-enhancing environment utilizing motivational gamified elements; music, exercise scenarios, visual or auditory feedback in order to provide a number of advantages for motivating behavior change. The user experiences the virtual environment through visual and audio feedback using a head-mounted device, flat screen, or projection system. It presents the opportunity for motor learning by testing the user's ability to solve problems and master real-world skills in a virtual environment by giving feedback. In considering all of the gamified features that are included in a rehabilitation program, it is important to ensure that they achieve the objectives of the rehabilitation program in which they are incorporated (validity).

Based on the recent published literatures, most of the studies that used different types of extended reality used devices utilised the Kinect camera or other devices that may not be affordable or easily accessible in terms of setting up to stroke survivors. To create real-world scenarios, the investigators have brought together the Exeter and Sao Paulo teams who have world-class expertise in developing VR software. The investigators intend to use some non-immersive VR adapted exercise scenarios with many levels of difficulties designed to be suitable and safe for home-based rehabilitation. The investigators have conducted a content validity and usability study with stroke survivors and physiotherapists aiming to refine these exercises to be more tailored and suitable to be delivered to stroke people at their homes. Based on this study, the investigators have found a good degree of agreement among the physiotherapist and stroke survivors regarding the suitability of these exercises for stroke home rehabilitation taking in consideration some suggestions to be more tailored according to patients' abilities. Based on these results, the investigators have created our newly adapted NOVEL program taking in considerations some important key features to be implemented in the newly developed exercises.

The overall aim of this mixed method feasibility RCT pilot study is to evaluate the feasibility and efficacy of a non-immersive VR home-based exercise program, compared to a usual care among stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Having stroke for more than 6 months (early or late chronic stage).
* Not participating in any other rehabilitation study.
* Able to read in English.
* Has good internet connection at home, or can the investigator give them a sim card.
* Score ≤2 on the Modified Ashworth Scale.
* Any degree of upper limb impairment due to stroke (Fugl-Meyer Assessment (FMA)-UE score <57).
* Having sufficient space at home.
* The participant should have a laptop, computer at their home, if they don't have any of that, the investigator can loan them a laptop.

Exclusion Criteria:

* Having severe arm, leg, or spine contractures, or deformities (MAS 3 or 4).
* Having any medical contraindications (seizure disorders, symptomatic shoulder subluxation, artificial cardiac pacemaker device, persistent shoulder pain (> 5 on VAS scale as an average).
* To ensure patients had sufficient cognitive abilities to participate in training and evaluation and to provide informed consent, the investigators will exclude patients diagnosed with - serious aphasia (cannot read the instructions) or cognitive dysfunction (inability to understand and follow two-stage instructions given by the investigators.
* To avoid potential confounding effects associated with other treatments, patients with any history of virtual reality upper-limb training or who received a botulinum toxin injection within 16 weeks before enrolment will be excluded.
* Insufficient motor control to move the avatar on the screen.
* Concurrent enrolment in another investigational study.
* Pregnancy (self reported).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible participants out of screened participants | During the screening process
  Total number of participants who pass the screening phase.
Proportion of ineligible participants out of screened patients | During the screening process
  Total number of participants who are ineligible with their reasons.
Success rate of obtaining consent from those eligible participants | During the enrolment process
  Number of participants enrolled/randomised
Retention rate of the participants | Recorded at week 8 at the end of delivering the intervention.
  Retention rate is defined as proportion of people that finished the exercise programme after 8 weeks. Retention data will be assessed based on (i) proportion of participants with complete outcome assessment; (ii) number of discontinuation and reasons.
Adherence of the participants | Recorded at week 8 at the end of delivering the intervention.
  Adherence is defined as the number and proportion of scheduled sessions undertaken by the participants.
Total number of adverse events reported by the participants using their workbook. | Recorded at week 8 at the end of delivering the intervention.
  Adverse events are any unfavourable experiences reported by participants during the study (regardless of whether these were related to the intervention). Participants in intervention and control groups will be asked to report any adverse events throughout the intervention period in their workbook and report any adverse effect to the researcher during the weekly meeting.

SECONDARY OUTCOMES:
Change from baseline in upper limb function on Fugl-Meyer Assessment for Upper Extremity (FMA-UE) test at week 8. | Completed at baseline and 8 weeks after receiving the intervention or the usual care.
  Fugl-Meyer Assessment for Upper Extremity (FMA-UE) is a valid tool to assess the upper limb motor function impairment among stroke survivors. The FMA-UE motor function score captures synergy, coordination, and sensorimotor functions (UE, wrist, and hand). The FMA-UE score has been shown to be valid in participants with stroke. This scale is one of the most widely used clinical scales for assessing upper extremity motor recovery after stroke, with 33 items, divided into 3 levels of scores, 0 (none), 1 (partial), and 2 (full)points respectively, according to the degree of task completion, and the total score was 66, with higher patient scores suggesting better motor function. FMA-UE is quantified by indicators and has the advantages of being detailed, reliable, and sensitive, which has been established as a standardized assessment tool to measure upper limb movement function.
Change from baseline in upper limb function on action research arm test (ARAT) at week 8. | Completed at baseline and 8 weeks after receiving the intervention or the usual care.
  ARAT (action research arm test) scale will be used to assess the upper limb functional impairment. It consists of 19 items focusing on grasping objects of different shapes and sizes, and gross arm movements. Each item is given an ordinal score of 0, 1, 2, or 3 with higher values indicating better function. The test has high inter-rater and test-retest reliability, good validity and is sensitive to therapy-related changes after stroke
Change from baseline in upper limb function on The Motor Activity Log test at week 8. | Completed at baseline and 8 weeks after receiving the intervention or the usual care.
  The Motor Activity Log is a valid and reliable self-report of quality of upper limb movement and amount of use, to capture the patient perspective. A clinically important mean change on the Motor Activity Log is ≥1; (scale range 0-5)
Change from baseline in balance confidence on Activities-Specific Balance Confidence(ABC) scale at week 8. | Completed at baseline and 8 weeks after receiving the intervention or the usual care.
  Regarding the balance confidence, The ABC scale, a 16-item structured questionnaire, will be used to measure participants' confidence in performing various activities without falling or feeling unsteady. The ABC score ranges from 0 (no confidence) to 100. the participant will rate each of the 16 items with a score ranging from 0% to 100%. after that, the total score will be divided by 16. Higher score means better balance confidence in doing the activities of daily living.
Change from baseline in trunk control on Trunk Impairment Scale (TIS) at week 8. | Completed at baseline and 8 weeks after receiving the intervention or the usual care.
  The trunk controls of the patients will be evaluated with the Trunk Impairment Scale (TIS). This scale evaluates the degree of motor loss in the trunk and trunk control in patients with stroke under the headings of static sitting balance, dynamic sitting balance and coordination. TIS consists of 17 items in total and each item is scored as 2 or 3 points. The total score is a minimum of 0 and a maximum of 23. High score indicates better trunk control. Test actions will be expressed verbally and visually by the researcher. TIS scoring will be done according to the performance of the patient.
Change from baseline in balance on Berg Balance Scale (BBS) at week 8. | Completed at baseline and 8 weeks after receiving the intervention or the usual care.
  The scale consists of 14 functional parameters that evaluate the static and dynamic balance in activities of daily living. The BBS assesses the ability to maintain balance during daily functional activities. Each parameter is scored between 0-4, with "0= unable to perform or requiring help," "4= normal performance." A higher score on the Berg Balance Scale indicates better balance. In the study, BBS assessment will be started with a sitting position. After activities such as sitting without support, getting up from a sitting position, the participant's balance will be observed in the standing position and with various activities. Adequate precautions will be considered against the risk of falling in the evaluation and the total score will be calculated according to the patient's performance.
User experience on User experience questionnaire (UEQ) at week 8. | Completed at week 8 after receiving the intervention.
  The UEQ assesses the patient experience after engaging in the original or modified NOVEL program. Each item of this questionnaire (a total of 26 items) of the UEQ consists of antonym-adjective pairs (e.g., annoying vs. enjoyable), which can be rated on a 7-point Likert scale ranging from-3(fully agree with a negative term) to+3 (fully agree with a positive term). They are randomly presented. The 26 items are grouped into six scales: attractiveness (general impression of the proposed game), perspicuity (how easy it is to get familiar with the proposed game), efficiency (solving tasks without unnecessary effort), dependability (feeling in control), stimulation (how exciting and motivating the proposed game is), and novelty (how innovative and creative the game is). This outcome measure will be used for the intervention groups 1 and 2 (no assessment for the control group as they are receiving the usual care).
Physical activity enjoyment on Physical activity enjoyment scale (PACES) at week 8. | Completed at week 8 after receiving the intervention.
  PACES is an 18-item scale that assesses the participants' enjoyment of the intervention they received. The participants are asked to rate how they felt about the NOVEL exercise program using a 7-point Likert scale from 1 (I enjoy it) to 7 (I hate it). PACES has 11 negatively worded items and 7 positively worded items. The scores range from 18 to 126, with a higher score indicating higher enjoyment. This outcome measure will be used for the intervention groups 1 and 2 (no assessment for the control group as they are receiving the usual care).
Change from baseline in quality of life on the EuroQol five-dimension scale (EQ-5D) at week 8. | Completed at baseline and 8 weeks after receiving the intervention or the usual care.
  The EuroQol five-dimension scale (EQ-5D) consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. This scale is a health status self-reporting scale designed to assess and value the health state and the quality of life across disease areas. It consists of 5 dimensions. Each dimension has 3 levels coded from 1 to 3: 1, no problems; 2, some problems; and 3, extreme problems. On each dimension, patients chose the answer that best described their health status, which resulted in a 5-number sequence describing each level of each dimension
Participant experience using semi-structured interviews at the end of receiving the intervention or the usual care. | completed after week 8.
  At the end of the study, the investigators are planning to do a qualitative semi-structured interviews with the participant in the experimental group aiming to understand stroke patients' experiences, facilitators and barriers after using the intervention. The interviews will be used to explore their experience of using the intervention or the usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Dawes, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No